CLINICAL TRIAL: NCT05838144
Title: Efficacy of Acapella on Spirometry Measures in Patients With Bronchiectasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-IMG-02/2023-505
Record Dates: First submitted 2023-03-24; First posted 2023-05-01 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acapella (Active Comparator): Will use Acapella device 3 times per day for 15 minutes for 7 days beside medications and routine physical therapy program.
  Interventions: Device: Acapella device; Other: Only routine chest physical therapy program
- Only routine physical therapy program (Placebo Comparator): Only they will receive medications and routine physical therapy program.
  Interventions: Other: Only routine chest physical therapy program

INTERVENTIONS:
Device: Acapella device — Group A. Will use Acapella device.
  Arms: Acapella
Other: Only routine chest physical therapy program — Group B. Will take medications and perform routine chest physical therapy program.

SUMMARY:
1. Acapella group. Will use Acapella device for 3 times per day for 15 minutes for 7 days beside medications and routine chest physical therapy program .
2. Only routine physical therapy program group ( control group). Will only take medications and routine chest physical therapy program.

DETAILED DESCRIPTION:
1. Acapella group.Will use Acapella device for 3 times per day for 15 minutes for 7 days beside medications and routine chest physical therapy program.
2. Only routine physical therapy program group( control group). Will only take medications and routine chest physical therapy program Spirometer measures such as forced vital capacity (FVC) and forced expiratory volume in the first second (FEV1) will be measured for every patient before and after the end of 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. bronchiectasis patients.
2. Age range between 40 to 55 years old of both gender.
3. Cooperative patients.

Exclusion Criteria:

1. Patients with severe cardiac disorders.
2. Un controlled hypertensive patients.
3. Un controlled diabetic patients.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Spirometry measures | 7 days
  FVC, FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Y Abo zaid, Principal Investigator — Lecturer
Locations (1):
- Shymaa yussuf abo zaid, Cairo, Egypt